CLINICAL TRIAL: NCT06681974
Title: RANDOMIZED CONTROLLED NON-INFERIORITY TRIAL TO ANALYZE THE EFFECTIVENESS OF OROPHARYNGEAL MYOFUNCTIONAL THERAPY IN MILD-MODERATE OBSTRUCTIVE SLEEP APNEA IN THE GENERAL POPULATION
Brief Title: OROPHARYNGEAL MYOFUNCTIONAL THERAPY IN OBSTRUCTIVE SLEEP APNEA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OMTOSA
Record Dates: First submitted 2024-07-17; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Oropharyngeal myofunctional therapy; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): indications on the hygienic-dietary measures
  Interventions: Behavioral: CONTROL:Information form with hygienic-dietary measures or sleep hygiene guidelines is provided and explained.
- experimental (Experimental): indications on the hygienic-dietary measures + an exercise program based on OMT for 20 weeks
  Interventions: Biological: EXPERIMENTAL: program of exercises that will be composed of 4 blocks

INTERVENTIONS:
Behavioral: CONTROL:Information form with hygienic-dietary measures or sleep hygiene guidelines is provided and explained. — * Establish a regular sleep schedule
  * Do not stay in bed longer than our regular sleep schedule.
  * Avoid naps during the day
  * Do not perform exciting activities and/or activities that demand physical or mental energy in the 3 hours prior to going to bed.
  * Avoid the use of mobile screens, as well as exposure to intense light in the 3 hours prior to going to bed.
  * Follow a healthy bedtime routine
  * Healthy lifestyle habits: avoid tobacco, alcohol and other toxic substances.
  Arms: control group
Biological: EXPERIMENTAL: program of exercises that will be composed of 4 blocks — the first is the work of the soft palate (retropalatine level), the second is the work of the functionality of the tongue (retroglossus level), the third is the work of the position of the hyoid bone (hypopharyngeal level), and the fourth is work on anterior head tilt and craniocervical extension (anterior head posture).
  Arms: experimental

SUMMARY:
Obstructive Sleep Apnea (OSA) is a prevalent nocturnal breathing disorder among the general population. Oropharyngeal myofunctional therapy (OMT) is an alternative conservative treatment used to improve OSA, associated health problems, and to improve the efficacy and tolerability of CPAP.

The objective is to determine the effect of OMT in the general population with mild-moderate OSA.

The overall study design will be a randomized controlled clinical trial with parallel groups. Both the control group and the intervention group will receive the same indications on the hygienic-dietary measures to be followed. The intervention group will also follow an exercise program based on OMT for 20 weeks. The effect on the apnea-hypopnea index and other variables will be determined by means of respiratory polygraphy before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance and signature of the informed consent
* Diagnosis of OSA with mild-moderate AHI without criteria for treatment with CPAP and/or other treatments (DAM).
* Patients who refused CPAP, were not candidates and/or refused DAM.
* Age > 18 years and < 70 years

Exclusion Criteria:

* Craniofacial malformations. Severe developmental delay. Intellectual disability.
* Diagnosis of neurodegenerative disease.
* Limited tongue mobility/presence of ankyloglossia as well as Temporo-Mandibular Joint pathology.
* Regular use of hypnotic medications
* Bulbar pathologies
* AHI of central origin above 50% of the total sleep time.
* Obesity grade II or more.
* Severe cardiovascular, neuromuscular or pulmonary pathology or chronic domiciliary oxygen use. Hypoventilation-obesity syndrome.
* Refuse to participate in the clinical trial despite fulfilling the inclusion criteria and not presenting any exclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
the effectiveness of Oropharyngeal myofunctional therapy in the treatment of Obstructive Sleep Apnea compared to conservative treatment measured by Respiratory Poligraphy | 12 months

SECONDARY OUTCOMES:
the effectiveness of Oropharyngeal myofunctional therapy in the treatment of Obstructive Sleep Apnea on nocturnal and diurnal clinical variable measured by means of the Epworth Test | 12 months
the impact of Oropharyngeal myofunctional therapy in Obstructive Sleep Apnea treatment on quality of life in the general population diagnosed with mild-moderate OSA using the EuroQol-5D questionnaire. | 12 months
the degree of tolerance of Oropharyngeal myofunctional therapy in patients diagnosed with mild-moderate Obstructive Sleep Apnea using a Likert-type design Visual Analog Scale Rating and Pairwise Comparison Rating Scale (VAS-RRP). | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital universitario Marques de Valdecilla, Santander, Spain

IPD SHARING:
Plan to Share IPD: No